CLINICAL TRIAL: NCT07105007
Title: Proof-of-concept of a Behavioral Intervention to Improve the Cardiovascular Health of People Living With HIV
Acronym: HEICA-HIV-2025
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); State University of Londrina (Other)
Responsible Party: Principal Investigator, Vitor Oliveira, Research Assistant Professor: School of Nursing., University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00022246
Record Dates: First submitted 2025-07-17; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: HIV; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single-arm pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicomponent (physical activity, education, behavioral coaching, mobile health) (Experimental): HEICA-HIV components will include: a) education sessions; b) exercise intervention; c) individual coaching; d) mobile health support. COMPONENT 1: Education Sessions. At the beginning of the program, the participants will receive two face-to-face group education sessions, consisting of 90 minutes of exercise and cardiovascular health education. COMPONENT 2: Exercise Intervention. After completing the education sessions, the participants will start 8 weeks of a hybrid exercise intervention, three days/week, being one supervised session in the exercise center and two unsupervised sessions at home. COMPONENT 3: Individual Coaching. At the end of their weekly in-person exercise sessions, the participants will receive a 20 min coaching session to address their attitudes, self-efficacy, and behavioral self-management skills towards exercise. COMPONENT 4: Mobile health support. At the beginning of the program, participants will receive a fitness activity tracker to help in achieving goals
  Interventions: Behavioral: Exercise Intervention; Behavioral: Education sessions; Behavioral: Behavioral coaching; Behavioral: Mobile health support

INTERVENTIONS:
Behavioral: Exercise Intervention — After completing the education sessions, the participants will start 8 weeks of a hybrid exercise intervention, three days/week, being one supervised session in the exercise center and two unsupervised sessions at home. Sessions at the exercise center will be supervised by experienced exercise trainers in a 1:1 ratio. The intervention is designed to meet the recommendation of at least 150 minutes of MVPA per week and the recommendations on exercise intensity and volume from the ACSM. Each exercise session will be composed of aerobic and resistance exercises at moderate intensity (i.e., combined exercise training), which is the best exercise model for the needs of PLWH. Additionally, poor muscle strength has been associated with lower VO2peak among PLWH, suggesting that appropriate muscle-strengthening exercises can improve the aerobic performance of these patients. The aerobic exercise will be performed in a continuous manner and prescribed using the heart rate reserve.
Behavioral: Education sessions — At the beginning of the program, the participants will receive two face-to-face group education sessions, consisting of 90 minutes of exercise and cardiovascular health education. The material for the education sessions will be developed by the study team (a diverse team including exercise scientists, nurse, cardiologist, and infectious disease specialist). The focus of the sessions will be to increase the participants' knowledge and self-efficacy. The education sessions will occur prior to the start of the exercise intervention, to teach the participants how to safely perform the home-based exercises. An interventionist, who will possess a degree in a health profession, will present the content following the completion of standard training using material and guidance developed for this purpose. The content of the sessions will include a self-assessment on exercise and physical activity, and incorporate the ACSM recommendations for quantity and quality of exercise
Behavioral: Behavioral coaching — At the end of their weekly in-person exercise sessions, the participants will receive a 20 minute coaching session to address their attitudes, self-efficacy, and behavioral self-management skills towards exercise. During the sessions, the trainers will be taught to use motivational interviewing, an evidence-based communication strategy that identifies and enhances patients' own motivations and reasons for health behavior change. Motivational interviewing is an approach to assessment and intervention based on the Stages of Motivational Readiness for Change model, which has been shown to increase physical activity in people with chronic health conditions. According to the Stages of Motivational Readiness for Change Model, individuals move through a series of stages (i.e., Precontemplation, Contemplation, Preparation, Action, and Maintenance) as they adopt and maintain a new habit. The coaching session will also address barriers from the home-based sessions, discuss HIV-specific barriers
Behavioral: Mobile health support — At the beginning of the program the participants will receive a fitness activity tracker (e.g., Fitbit or similar) to help in achieving their PA goals. Contemporary activity trackers provide reliable information on heart rate, steps count, and amount of PA performed, that will help the participants to monitor the intensity and amount during the home-base sessions. Heart rate monitoring will also be used to assess compliance with the home-based exercise prescription. Trackers also include gamification, awarding badges and trophies when goals are attained, that is demonstrated to be motivating.

SUMMARY:
Heart failure (HF) is a growing health and economic burden around the globe, and it remains a leading cause of morbidity and mortality among the general population. HIV is recognized as an independent risk factor for HF, due to direct and indirect effects. Furthermore, people living with HIV (PLWH) now have an increased life expectancy due to the evolution and widespread use of antiretroviral therapy (ART), leading to a rising burden of cardiovascular disease (CVD) and HF among this population. Yet, the provision of appropriate guideline-recommended cardiovascular care is lower in PLWH compared to the general population, and there are no studies testing HF prevention interventions focused on PLWH. Current guidelines for HF management highlight the importance of a healthy lifestyle in preventing and treating HF. Among PLWH, tailored, innovative, and sustainable exercise delivery models are necessary to overcome barriers and increase physical activity (PA) adherence in this population.

Building on the research team's prior mixed methods work and research expertise on exercise trials for PLWH, the investigators propose the Hybrid Exercise Intervention for Cardiovascular Health of People living with HIV (HEICA-HIV). HEICA-HIV is a novel multi-component 8-week intervention that will simultaneously deliver a supervised center-based (once a week) and a tailored home-based (twice a week) exercise intervention, together with exercise and cardiovascular health education. It will also involve behavioral coaching and mobile health support. The investigators evidence suggests that, by providing weekly exercise supervision together with a home-based prescription, the investigators can overcome difficulties associated with home-based programs (e.g., less intensive exercise training, less social support, and less face-to-face monitoring), and still observe the augmented health benefits obtained from supervised programs. Additionally, by requiring less time at the training center, this hybrid model can help with time restraints and transportation issues affecting marginalized populations, potentially increasing long-term exercise adherence in those who need it most. In this initial stage, HEICA-HIV will be focused on improving time in moderate-to-vigorous physical activity (MVPA). International guidelines recommend that every adult should engage in at least 150 minutes of MVPA per week in order to achieve optimal health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection (verified on medical record)
* Age ≥40 years
* Classified as heart failure stage A or B (American Heart Association Guidelines)
* On antiretroviral therapy (ART) for ≥12 months
* HIV RNA <200 copies/mL in the past 12 months
* Not engaged in a structured exercise or weight loss program in the past 6 months
* Physically inactive, defined as an activity level of less than 400 METs measured with the Global Physical Activity Questionnaire (GPAQ)
* Independent in basic activities of daily living
* Able to ambulate independently

Exclusion Criteria:

* Heart failure stage C or D (AHA Guidelines)
* Participating in structured exercise or weight loss program in the past 6 months
* BMI <18 or >48
* Exercising ≥3 times per week (≥20 minutes per session)
* Use of GLP-1 or other weight loss medications, or weight loss surgery within 6 months prior to enrollment
* Do not report fatigue
* Significant comorbidities (e.g., uncontrolled hypertension, severe musculoskeletal/neurological conditions)
* Inability to undergo MRI safely
* Pregnant or postmenopausal women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Adherence | From enrollment to the end of treatment at 8 weeks
  Description: Number of exercise and education sessions attended by each participant during the intervention.
  Unit of Measure: Number of sessions attended
Time Spent in Sedentary Behavior | From enrollment to the end of treatment at 8 weeks
  Description: Exploratory analysis of the average time spent in sedentary behavior per week.
  Unit of Measure: Minutes per week
Daily Step Count | From enrollment to the end of treatment at 8 weeks
  Description: Exploratory outcome assessing the average daily number of steps. Unit of Measure: Steps per day
Moderate to Vigorous Physical Activity (MVPA) Time | From enrollment to the end of treatment at 8 weeks
  Description: The primary outcome will be the objectively measured amount of time (in minutes) spent in moderate to vigorous physical activity (MVPA) per week.
  Assessment Method: Using the wGT3X-BT ActiGraph accelerometer (ActiGraph, LLC, Fort Walton Beach, FL), participants will wear the device for 7 consecutive days during waking hours. Data will be considered valid with at least 10 hours/day of wear time for at least 4 days.
  Data Processing: Data will be reduced using ActiLife software and MVPA will be classified based on Sasaki et al. adult cutpoints.
  Unit of Measure: Minutes per week

SECONDARY OUTCOMES:
High-sensitivity C-reactive Protein (hs-CRP) | From enrollment to the end of treatment at 8 weeks
  Description: Change in serum levels of hs-CRP from baseline to end of intervention.
  Unit of Measure: mg/L
B-type Natriuretic Peptide (BNP) | From enrollment to the end of treatment at 8 weeks
  Description: Change in serum levels of BNP from baseline to end of intervention.
  Unit of Measure: pg/mL
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | From enrollment to the end of treatment at 8 weeks
  Description: Change in serum levels of NT-proBNP from baseline to end of intervention.
  Unit of Measure: pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Oliveira, PhD, Principal Investigator — University of Washington
Locations (2):
- University of Washington, Seattle, Washington, United States
- Londrina State University, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No